CLINICAL TRIAL: NCT02162459
Title: Strength-enhancing Effect of Whey Protein Supplementation Following Resistance Exercise in Adolescent Males
Status: Completed | Type: Observational
Sponsor: Olympia Eye Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 1 dated January 2014
Record Dates: First submitted 2014-06-09; First posted 2014-06-12 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: Adolescent; supplements; strength; whey protein; bench press strength; squat strength

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- whey beverage: consumption of 52 grams of whey protein supplement following resistance exercise
- chocolate milk beverage: consumption of chocolate flavored milk following resistance exercise

SUMMARY:
This study investigates the strength gains associated with resistance training in a group of 18 male high school athletes consuming either a whey protein supplement or chocolate milk following their exercise.

ELIGIBILITY:
Inclusion Criteria:

* member of Bellarmine Preparatory School boys sports team
* Must be willing to consume a post-exercise beverage

Exclusion Criteria:

* allergy to either beverage

Ages: 16 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: male high school athletes
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
bench press strength | 8 weeks
  Calculated 1-repetition maximum bench press strength

SECONDARY OUTCOMES:
squat strength | 8 weeks
  calculated 1-repetition squat strength

CONTACTS AND LOCATIONS:
Overall Officials: Rodger D Bodoia, M.D., Study Chair — Olympia Eye Clinic
Locations (1):
- Bellarmine Preparatory School, Tacoma, Washington, United States